CLINICAL TRIAL: NCT03496298
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Effect of Efpeglenatide on Cardiovascular Outcomes in Type 2 Diabetes Patients at High Cardiovascular Risk
Brief Title: Effect of Efpeglenatide on Cardiovascular Outcomes
Acronym: AMPLITUDE-O
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to cancel TRIAL, not related to safety concern
Sponsor: Sanofi (Industry)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC14828; 2017-002954-35 (EudraCT Number); U1111-1186-2533 (Other: UTN)
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — efpeglenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo (matched to Efpeglenatide) as subcutaneous (SC) injection once weekly up to end of treatment.
  Interventions: Drug: Placebo
- Efpeglenatide 4 mg (Experimental): Participants received Efpeglenatide as SC injection 2 milligrams (mg) per week for 4 weeks then 4 mg per week up to end of treatment.
  Interventions: Drug: Efpeglenatide (SAR439977)
- Efpeglenatide 6 mg (Experimental): Participants received Efpeglenatide as SC injection 2 mg per week for 4 weeks, then 4 mg per week for 4 weeks and then 6 mg per week up to end of treatment.
  Interventions: Drug: Efpeglenatide (SAR439977)

INTERVENTIONS:
Drug: Efpeglenatide (SAR439977) — Pharmaceutical form: Solution for injection,
  Route of administration: SC
  Arms: Efpeglenatide 4 mg; Efpeglenatide 6 mg
Drug: Placebo — Pharmaceutical form: Solution for injection
  Route of administration: SC
  Arms: Placebo

SUMMARY:
Primary Objective:

To demonstrate that efpeglenatide 4 and 6 mg was noninferior to placebo on 3-point major adverse cardiac events (MACE) in Type 2 diabetes mellitus (T2DM) participants at high cardiovascular (CV) risk.

Secondary Objectives:

To demonstrate that efpeglenatide 4 and 6 mg was superior to placebo in T2DM participants with high CV risk on the following parameters:

* 3-point MACE.
* Expanded CV outcome.
* Composite outcome of new or worsening nephropathy.

To assess the safety and tolerability of efpeglenatide 4 and 6 mg, both added to standard of care in T2DM participants at high CV risk.

DETAILED DESCRIPTION:
The study duration per participant was up to approximately 36 months.

ELIGIBILITY:
Inclusion criteria:

* T2DM with glycosylated hemoglobin (HbA1c) greater than (>) 7 percentage.
* Age 18 years or older who met at least one of the cardiovascular disease criteria or age 50 years (male), 55 years (female) or older with glomerular filtration rate greater than or equal to 25 and less than 60 milliliters per minute and at least had one cardiovascular risk factor.
* Female participants agreed to follow contraceptive guidance.
* Signed written informed consent.

Exclusion criteria:

* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting.
* History of chronic pancreatitis or acute idiopathic pancreatitis or diagnosis of any type of acute pancreatitis within 3 months prior to screening.
* Personal or family history of medullary thyroid cancer.
* Hypertension (with a systolic blood pressure >180 millimeters of Mercury [mmHg] and/or diastolic blood pressure >100 mmHg).
* Hospitalization for hypertensive emergency within 3 months prior to randomization.
* Planned coronary procedure or surgery after randomization.
* No documented ophthalmologic exam with fundoscopy within 6 months prior to randomization.
* Retinopathy or maculopathy with treatment, either recent (3 months prior to randomization) or planned during the study.
* Treated with any glucagon-like peptide-1 receptor agonist product alone (eg, exenatide, liraglutide, lixisenatide, albiglutide, dulaglutide, semaglutide) or in combination within 3 months prior to screening.
* Use of any Dipeptidyl peptidase 4 inhibitor within 3 months prior to screening.
* Antihyperglycemic treatment had not been stable within 3 months prior to screening.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4076 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (353):
- United States (79):
  - Investigational Site Number 8400032, Sheffield, Alabama
  - Investigational Site Number 8400014, Gilbert, Arizona
  - Investigational Site Number 8400012, Surprise, Arizona
  - Investigational Site Number 8400046, Tucson, Arizona
  - Investigational Site Number 8400022, Beverly Hills, California
  - Investigational Site Number 8400065, Concord, California
  - Investigational Site Number 8400060, Greenbrae, California
  - Investigational Site Number 8400084, Long Beach, California
  - Investigational Site Number 8400002, Los Gatos, California
  - Investigational Site Number 8400085, Northridge, California
  - Investigational Site Number 8400082, Pomona, California
  - Investigational Site Number 8400025, Sacramento, California
  - Investigational Site Number 8400064, Englewood, Colorado
  - Investigational Site Number 8400019, Hamden, Connecticut
  - Investigational Site Number 8400023, Waterbury, Connecticut
  - Investigational Site Number 8400091, Hialeah, Florida
  - Investigational Site Number 8400040, Hollywood, Florida
  - Investigational Site Number 8400073, Hudson, Florida
  - Investigational Site Number 8400011, Jacksonville, Florida
  - Investigational Site Number 8400017, Jacksonville, Florida
  - Investigational Site Number 8400042, Jacksonville, Florida
  - Investigational Site Number 8400027, Miami, Florida
  - Investigational Site Number 8400051, Miami, Florida
  - Investigational Site Number 8400041, New Port Richey, Florida
  - Investigational Site Number 8400059, Ormond Beach, Florida
  - Investigational Site Number 8400006, Macon, Georgia
  - Investigational Site Number 8400008, Roswell, Georgia
  - Investigational Site Number 8400081, Idaho Falls, Idaho
  - Investigational Site Number 8400095, Arlington Heights, Illinois
  - Investigational Site Number 8400070, Chicago, Illinois
  - Investigational Site Number 8400036, Crystal Lake, Illinois
  - Investigational Site Number 8400030, New Albany, Indiana
  - Investigational Site Number 8400074, Topeka, Kansas
  - Investigational Site Number 8400077, Owensboro, Kentucky
  - Investigational Site Number 8400043, Paris, Kentucky
  - Investigational Site Number 8400034, Alexandria, Louisiana
  - Investigational Site Number 8400079, Monroe, Louisiana
  - Investigational Site Number 8400013, New Orleans, Louisiana
  - Investigational Site Number 8400047, Oxon Hill, Maryland
  - Investigational Site Number 8400001, Flint, Michigan
  - Investigational Site Number 8400061, Flint, Michigan
  - Investigational Site Number 8400010, Troy, Michigan
  - Investigational Site Number 8400005, Troy, Michigan
  - Investigational Site Number 8400024, Saint Paul, Minnesota
  - Investigational Site Number 8400045, St Louis, Missouri
  - Investigational Site Number 8400071, Billings, Montana
  - Investigational Site Number 8400028, Great Falls, Montana
  - Investigational Site Number 8400086, Kalispell, Montana
  - Investigational Site Number 8400037, Las Vegas, Nevada
  - Investigational Site Number 8400087, Raritan, New Jersey
  - Investigational Site Number 8400056, Staten Island, New York
  - Investigational Site Number 8400018, The Bronx, New York
  - Investigational Site Number 8400076, Greenville, North Carolina
  - Investigational Site Number 8400007, Morehead City, North Carolina
  - Investigational Site Number 8400093, Morehead City, North Carolina
  - Investigational Site Number 8400094, Morganton, North Carolina
  - Investigational Site Number 8400029, Fargo, North Dakota
  - Investigational Site Number 8400031, Columbus, Ohio
  - Investigational Site Number 8400078, Lorain, Ohio
  - Investigational Site Number 8400072, Bend, Oregon
  - Investigational Site Number 8400067, Beaver, Pennsylvania
  - Investigational Site Number 8400096, Philadelphia, Pennsylvania
  - Investigational Site Number 8400021, Pittsburgh, Pennsylvania
  - Investigational Site Number 8400015, Greer, South Carolina
  - Investigational Site Number 8400063, Murrells Inlet, South Carolina
  - Investigational Site Number 8400044, Rapid City, South Dakota
  - Investigational Site Number 8400016, Memphis, Tennessee
  - Investigational Site Number 8400009, Nashville, Tennessee
  - Investigational Site Number 8400055, Corpus Christi, Texas
  - Investigational Site Number 8400097, Dallas, Texas
  - Investigational Site Number 8400088, El Paso, Texas
  - Investigational Site Number 8400058, Fort Worth, Texas
  - Investigational Site Number 8400069, Houston, Texas
  - Investigational Site Number 8400089, Houston, Texas
  - Investigational Site Number 8400092, Richmond, Texas
  - Investigational Site Number 8400033, Waco, Texas
  - Investigational Site Number 8400039, Salt Lake City, Utah
  - Investigational Site Number 8400052, Norfolk, Virginia
  - Investigational Site Number 8400049, Manitowoc, Wisconsin
- Argentina (18):
  - Investigational Site Number 0320009, Buenos Aires
  - Investigational Site Number 0320002, Caba
  - Investigational Site Number 0320013, Caba
  - Investigational Site Number 0320010, Caba
  - Investigational Site Number 0320005, Caba
  - Investigational Site Number 0320008, Capital Federal
  - Investigational Site Number 0320001, Capital Federal
  - Investigational Site Number 0320004, Corrientes
  - Investigational Site Number 0320012, Corrientes
  - Investigational Site Number 0320011, Godoy Cruz
  - Investigational Site Number 0320007, Mar del Plata
  - Investigational Site Number 0320006, Merlo
  - Investigational Site Number 0320015, Rosario
  - Investigational Site Number 0320017, Rosario
  - Investigational Site Number 0320003, Salta
  - Investigational Site Number 0320018, Salta
  - Investigational Site Number 0320016, San Isidro
  - Investigational Site Number 0320014, Santa Rosa
- Bulgaria (15):
  - Investigational Site Number 1000011, Blagoevgrad
  - Investigational Site Number 1000014, Dimitrovgrad
  - Investigational Site Number 1000017, Gabrovo
  - Investigational Site Number 1000007, Kazanlak
  - Investigational Site Number 1000013, Kyustendil
  - Investigational Site Number 1000010, Lovech
  - Investigational Site Number 1000008, Plovdiv
  - Investigational Site Number 1000002, Plovdiv
  - Investigational Site Number 1000012, Rousse
  - Investigational Site Number 1000003, Sofia
  - Investigational Site Number 1000001, Sofia
  - Investigational Site Number 1000005, Sofia
  - Investigational Site Number 1000006, Stara Zagora
  - Investigational Site Number 1000009, Varna
  - Investigational Site Number 1000016, Yambol
- Canada (31):
  - Investigational Site Number 1240001, Barrie
  - Investigational Site Number 1240002, Brampton
  - Investigational Site Number 1240018, Burlington
  - Investigational Site Number 1240021, Burlington
  - Investigational Site Number 1240007, Calgary
  - Investigational Site Number 1240020, Calgary
  - Investigational Site Number 1240024, Chicoutimi
  - Investigational Site Number 1240004, Concord
  - Investigational Site Number 1240005, Etobicoke
  - Investigational Site Number 1240022, Greater Sudbury
  - Investigational Site Number 1240011, Lévis
  - Investigational Site Number 1240025, London
  - Investigational Site Number 1240028, London
  - Investigational Site Number 1240029, Mirabel
  - Investigational Site Number 1240008, Montreal
  - Investigational Site Number 1240031, Montreal
  - Investigational Site Number 1240014, Montreal
  - Investigational Site Number 1240023, Montreal
  - Investigational Site Number 1240017, Montreal
  - Investigational Site Number 1240015, Oakville
  - Investigational Site Number 1240012, Oshawa
  - Investigational Site Number 1240030, Ottawa
  - Investigational Site Number 1240027, Peterborough
  - Investigational Site Number 1240016, Pointe-Claire
  - Investigational Site Number 1240010, Québec
  - Investigational Site Number 1240019, Red Deer
  - Investigational Site Number 1240006, Sherbrooke
  - Investigational Site Number 1240013, Toronto
  - Investigational Site Number 1240003, Vancouver
  - Investigational Site Number 1240026, Victoria
  - Investigational Site Number 1240009, Victoriaville
- Chile (13):
  - Investigational Site Number 1520012, Antofagasta
  - Investigational Site Number 1520008, Concepción
  - Investigational Site Number 1520013, Santiago
  - Investigational Site Number 1520002, Santiago
  - Investigational Site Number 1520007, Santiago
  - Investigational Site Number 1520011, Santiago
  - Investigational Site Number 1520010, Santiago
  - Investigational Site Number 1520001, Santiago
  - Investigational Site Number 1520003, Santiago
  - Investigational Site Number 1520014, Santiago
  - Investigational Site Number 1520005, Santiago
  - Investigational Site Number 1520006, Temuco
  - Investigational Site Number 1520004, Viña del Mar
- Denmark (5):
  - Investigational Site Number 2080004, Aarhus N
  - Investigational Site Number 2080005, Esbjerg
  - Investigational Site Number 2080001, Hellerup
  - Investigational Site Number 2080003, Hvidovre
  - Investigational Site Number 2080002, København NV
- Estonia (3):
  - Investigational Site Number 2330002, Pärnu
  - Investigational Site Number 2330001, Tallinn
  - Investigational Site Number 2330003, Viljandi
- Finland (4):
  - Investigational Site Number 2460002, Helsinki
  - Investigational Site Number 2460001, Jyväskylä
  - Investigational Site Number 2460003, Kuopio
  - Investigational Site Number 2460004, Oulu
- Germany (8):
  - Investigational Site Number 2760006, Berlin
  - Investigational Site Number 2760009, Berlin
  - Investigational Site Number 2760004, Essen
  - Investigational Site Number 2760008, Frankfurt am Main
  - Investigational Site Number 2760005, Münster
  - Investigational Site Number 2760003, Oldenburg in Holstein
  - Investigational Site Number 2760002, Pirna
  - Investigational Site Number 2760007, Rotenburg an der Fulda
- Hungary (11):
  - Investigational Site Number 3480012, Balatonfüred
  - Investigational Site Number 3480011, Budapest
  - Investigational Site Number 3480003, Budapest
  - Investigational Site Number 3480005, Budapest
  - Investigational Site Number 3480001, Budapest
  - Investigational Site Number 3480006, Budapest
  - Investigational Site Number 3480002, Debrecen
  - Investigational Site Number 3480009, Komárom
  - Investigational Site Number 3480008, Mosonmagyaróvár
  - Investigational Site Number 3480007, Székesfehérvár
  - Investigational Site Number 3480004, Zalaegerszeg
- India (9):
  - Investigational Site Number 3560001, Belagavi
  - Investigational Site Number 3560002, Gūrgaon
  - Investigational Site Number 3560007, Kolkata
  - Investigational Site Number 3560006, Lucknow
  - Investigational Site Number 3560003, New Delhi
  - Investigational Site Number 3560009, New Delhi
  - Investigational Site Number 3560010, Pune
  - Investigational Site Number 3560005, Pune
  - Investigational Site Number 3560004, Vellore
- Italy (6):
  - Investigational Site Number 3800006, Catania
  - Investigational Site Number 3800003, Catanzaro
  - Investigational Site Number 3800005, Catanzaro
  - Investigational Site Number 3800002, Chieti
  - Investigational Site Number 3800001, Milan
  - Investigational Site Number 3800004, Roma
- Latvia (4):
  - Investigational Site Number 4280004, Daugavpils
  - Investigational Site Number 4280002, Liepāja
  - Investigational Site Number 4280001, Riga
  - Investigational Site Number 4280003, Sigulda
- Lithuania (4):
  - Investigational Site Number 4400001, Kaunas
  - Investigational Site Number 4400002, Kaunas
  - Investigational Site Number 4400003, Klaipėda
  - Investigational Site Number 4400004, Vilnius
- Mexico (14):
  - Investigational Site Number 4840004, Actopan
  - Investigational Site Number 4840007, Aguascalientes
  - Investigational Site Number 4840009, Aguascalientes
  - Investigational Site Number 4840013, Aguascalientes
  - Investigational Site Number 4840014, Chihuahua City
  - Investigational Site Number 4840002, Cuernavaca
  - Investigational Site Number 4840016, Durango
  - Investigational Site Number 4840015, Durango
  - Investigational Site Number 4840006, Guadalajara
  - Investigational Site Number 4840003, Guadalajara
  - Investigational Site Number 4840005, Guadalajara
  - Investigational Site Number 4840011, Monterrey
  - Investigational Site Number 4840010, Monterrey
  - Investigational Site Number 4840001, Monterrey
- Norway (3):
  - Investigational Site Number 5780002, Hamar
  - Investigational Site Number 5780001, Oslo
  - Investigational Site Number 5780003, Stavanger
- Peru (7):
  - Investigational Site Number 6040007, Lima
  - Investigational Site Number 6040004, Lima
  - Investigational Site Number 6040003, Lima
  - Investigational Site Number 6040006, Lima
  - Investigational Site Number 6040001, Lima
  - Investigational Site Number 6040005, Lima
  - Investigational Site Number 6040002, Piura
- Poland (15):
  - Investigational Site Number 6160017, Bialystok
  - Investigational Site Number 6160018, Bydgoszcz
  - Investigational Site Number 6160015, Bydgoszcz
  - Investigational Site Number 6160016, Gdansk
  - Investigational Site Number 6160012, Gdansk
  - Investigational Site Number 6160005, Katowice
  - Investigational Site Number 6160006, Płock
  - Investigational Site Number 6160011, Skierniewice
  - Investigational Site Number 6160013, Skorzewo
  - Investigational Site Number 6160010, Szczecin
  - Investigational Site Number 6160007, Torun
  - Investigational Site Number 6160009, Torun
  - Investigational Site Number 6160014, Tychy
  - Investigational Site Number 6160002, Warsaw
  - Investigational Site Number 6160004, Wroclaw
- Romania (10):
  - Investigational Site Number 6420007, Bacau
  - Investigational Site Number 6420001, Brasov
  - Investigational Site Number 6420011, Brasov
  - Investigational Site Number 6420009, Bucharest
  - Investigational Site Number 6420012, Oradea
  - Investigational Site Number 6420005, Oradea
  - Investigational Site Number 6420010, Oradea
  - Investigational Site Number 6420008, Ploieşti
  - Investigational Site Number 6420002, Târgu Mureş
  - Investigational Site Number 6420003, Târgu Mureş
- Russia (18):
  - Investigational Site Number 6430018, Kaliningrad
  - Investigational Site Number 6430014, Kazan'
  - Investigational Site Number 6430001, Kemerovo
  - Investigational Site Number 6430017, Krasnogorsk
  - Investigational Site Number 6430004, Moscow
  - Investigational Site Number 6430005, Moscow
  - Investigational Site Number 6430002, Moscow
  - Investigational Site Number 6430015, Moscow
  - Investigational Site Number 6430009, Novosibirsk
  - Investigational Site Number 6430019, Novosibirsk
  - Investigational Site Number 6430006, Saint Petersburg
  - Investigational Site Number 6430010, Saint Petersburg
  - Investigational Site Number 6430011, Saint Petersburg
  - Investigational Site Number 6430013, Saint Petersburg
  - Investigational Site Number 6430016, Saint Petersburg
  - Investigational Site Number 6430012, Saint Petersburg
  - Investigational Site Number 6430003, Saratov
  - Investigational Site Number 6430020, Saratov
- Serbia (6):
  - Investigational Site Number 6880001, Belgrade
  - Investigational Site Number 6880002, Belgrade
  - Investigational Site Number 6880003, Belgrade
  - Investigational Site Number 6880005, Belgrade
  - Investigational Site Number 6880004, Kragujevac
  - Investigational Site Number 6880006, Novi Sad
- Slovakia (12):
  - Investigational Site Number 7030007, Bratislava
  - Investigational Site Number 7030001, Košice
  - Investigational Site Number 7030004, Košice
  - Investigational Site Number 7030003, Kráľovský Chlmec
  - Investigational Site Number 7030009, Moldava nad Bodvou
  - Investigational Site Number 7030010, Pezinok
  - Investigational Site Number 7030006, Považská Bystrica
  - Investigational Site Number 7030005, Prešov
  - Investigational Site Number 7030008, Rožňava
  - Investigational Site Number 7030011, Štúrovo
  - Investigational Site Number 7030002, Trebišov
  - Investigational Site Number 7030012, Trenčín
- South Africa (8):
  - Investigational Site Number 7100007, Bloemfontein
  - Investigational Site Number 7100005, Cape Town
  - Investigational Site Number 7100006, Cape Town
  - Investigational Site Number 7100003, Johannesburg
  - Investigational Site Number 7100001, Johannesburg
  - Investigational Site Number 7100002, Parow
  - Investigational Site Number 7100004, Rivonia
  - Investigational Site Number 7100008, Umhlanga Rocks Suburb
- South Korea (10):
  - Investigational Site Number 4100006, Guri-si, Gyeonggi-do
  - Investigational Site Number 4100007, Busan
  - Investigational Site Number 4100005, Seoul
  - Investigational Site Number 4100002, Seoul
  - Investigational Site Number 4100009, Seoul
  - Investigational Site Number 4100001, Seoul
  - Investigational Site Number 4100011, Seoul
  - Investigational Site Number 4100003, Seoul
  - Investigational Site Number 4100010, Seoul
  - Investigational Site Number 4100008, Wŏnju
- Spain (13):
  - Investigational Site Number 7240008, Alcorcón
  - Investigational Site Number 7240002, Barcelona
  - Investigational Site Number 7240009, Barcelona
  - Investigational Site Number 7240007, Granada
  - Investigational Site Number 7240010, Madrid
  - Investigational Site Number 7240001, Madrid
  - Investigational Site Number 7240006, Majadahonda
  - Investigational Site Number 7240011, Málaga
  - Investigational Site Number 7240005, Olot
  - Investigational Site Number 7240003, San Sebastián de los Reyes
  - Investigational Site Number 7240013, Seville
  - Investigational Site Number 7240004, Valencia
  - Investigational Site Number 7240014, Valencia
- Sweden (6):
  - Investigational Site Number 7520006, Gothenburg
  - Investigational Site Number 7520003, Helsingborg
  - Investigational Site Number 7520004, Kristianstad
  - Investigational Site Number 7520002, Malmo
  - Investigational Site Number 7520005, Skövde
  - Investigational Site Number 7520001, Stockholm
- Turkey (Türkiye) (12):
  - Investigational Site Number 7920005, Adana
  - Investigational Site Number 7920010, Ankara
  - Investigational Site Number 7920012, Antalya
  - Investigational Site Number 7920015, Aydin
  - Investigational Site Number 7920002, Bursa
  - Investigational Site Number 7920013, Eskişehir
  - Investigational Site Number 7920001, Istanbul
  - Investigational Site Number 7920006, Istanbul
  - Investigational Site Number 7920011, İzmit
  - Investigational Site Number 7920014, Kütahya
  - Investigational Site Number 7920007, Samsun
  - Investigational Site Number 7920009, Sivas
- Ukraine (9):
  - Investigational Site Number 8040006, Dnipro
  - Investigational Site Number 8040009, Ivano-Frankivsk
  - Investigational Site Number 8040001, Ivano-Frankivsk
  - Investigational Site Number 8040003, Kharkiv
  - Investigational Site Number 8040002, Kharkiv
  - Investigational Site Number 8040007, Kiev
  - Investigational Site Number 8040008, Kyiv
  - Investigational Site Number 8040004, Ternopil
  - Investigational Site Number 8040005, Vinnytsia

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) by Sanofi: product rights transferred to Hanmi pharmaceutical.

REFERENCES:
- [Result] Gerstein HC, Sattar N, Rosenstock J, Ramasundarahettige C, Pratley R, Lopes RD, Lam CSP, Khurmi NS, Heenan L, Del Prato S, Dyal L, Branch K; AMPLITUDE-O Trial Investigators. Cardiovascular and Renal Outcomes with Efpeglenatide in Type 2 Diabetes. N Engl J Med. 2021 Sep 2;385(10):896-907. doi: 10.1056/NEJMoa2108269. Epub 2021 Jun 28. PMID 34215025
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Gerstein HC, Li Z, Ramasundarahettige C, Baek S, Branch KRH, Del Prato S, Lam CSP, Lopes RD, Pratley R, Rosenstock J, Sattar N. Exploring the Relationship Between Efpeglenatide Dose and Cardiovascular Outcomes in Type 2 Diabetes: Insights From the AMPLITUDE-O Trial. Circulation. 2023 Mar 28;147(13):1004-1013. doi: 10.1161/CIRCULATIONAHA.122.063716. Epub 2023 Feb 20. PMID 36802715
- [Derived] Lam CSP, Ramasundarahettige C, Branch KRH, Sattar N, Rosenstock J, Pratley R, Del Prato S, Lopes RD, Niemoeller E, Khurmi NS, Baek S, Gerstein HC. Efpeglenatide and Clinical Outcomes With and Without Concomitant Sodium-Glucose Cotransporter-2 Inhibition Use in Type 2 Diabetes: Exploratory Analysis of the AMPLITUDE-O Trial. Circulation. 2022 Feb 22;145(8):565-574. doi: 10.1161/CIRCULATIONAHA.121.057934. Epub 2021 Nov 14. PMID 34775781
- [Derived] Gerstein HC, Branch K, Heenan L, Del Prato S, Khurmi NS, Lam CSP, Pratley R, Rosenstock J, Sattar N. Design and baseline characteristics of the AMPLITUDE-O cardiovascular outcomes trial of efpeglenatide, a weekly glucagon-like peptide-1 receptor agonist. Diabetes Obes Metab. 2021 Feb;23(2):318-323. doi: 10.1111/dom.14223. Epub 2020 Oct 22. PMID 33026143

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 344 active sites in 28 countries. Overall, 5732 participants were screened between 27 April 2018 and 25 April 2019; of whom 4076 participants were randomized by interactive response technology (1:1:1 ratio) to receive placebo, efpeglenatide 4 milligrams (mg) or efpeglenatide 6 mg. Screen failures were mainly due to inclusion criteria not met.
Pre-assignment Details: Randomization was stratified by the current or potential future use of a sodium-glucose co-transporter-2 (SGLT2) inhibitor: current use; potential future use; neither current nor potential future use.
Groups:
- Placebo: Participants received placebo (matched to Efpeglenatide) as subcutaneous (SC) injection once weekly up to end of treatment (median duration: 19.8 months).
- Efpeglenatide 4 mg: Participants received Efpeglenatide as SC injection 2 mg per week for 4 weeks then 4 mg per week up to end of treatment (median duration: 19.9 months).
- Efpeglenatide 6 mg: Participants received Efpeglenatide as SC injection 2 mg per week for 4 weeks, then 4 mg per week for 4 weeks and then 6 mg per week up to end of treatment (median duration: 20 months).
Period: Overall Study
Arm/Group | Placebo | Efpeglenatide 4 mg | Efpeglenatide 6 mg
Started (Randomized.) | 1359 | 1359 | 1358
Randomized and Treated | 1358 | 1358 | 1357
Safety Population (Safety population included all randomized participants who had received at least 1 dose of double-blind treatment, regardless of the amount of treatment administered and were analyzed according to treatment actually received.) | 1355 (2 participants of Placebo arm received Efpeglenatide 4 mg treatment and 1 participant received Efpeglenatide 6 mg treatment. Hence, they were counted in the respective arm for safety analysis.) | 1360 (2 participants of Placebo arm received Efpeglenatide 4 mg treatment and thus counted in the 4 mg treatment arm for safety analysis.) | 1358 (1 participant of Placebo arm received Efpeglenatide 6 mg treatment and thus counted in the 6 mg treatment arm for safety analysis.)
Completed | 42 | 36 | 23
Not Completed | 1317 | 1323 | 1335
Not completed — Adverse Event | 49 | 68 | 79
Not completed — Study terminated by Sponsor | 1050 | 1063 | 1071
Not completed — Physician decision (other than Adverse event) | 12 | 17 | 10
Not completed — Withdrawal by Subject | 176 | 154 | 151
Not completed — Other | 29 | 20 | 23
Not completed — Randomized and not treated | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent-to-treat (ITT) population that included all randomized participants irrespective of compliance with the study protocol and procedures and were analyzed in the treatment group to which they were randomized.
Groups:
- Placebo: Participants received placebo (matched to Efpeglenatide) as SC injection once weekly up to end of treatment (median duration: 19.8 months).
- Total: Total of all reporting groups
Arm/Group | Placebo | Efpeglenatide 4 mg | Efpeglenatide 6 mg | Total
Number analyzed (Participants) | 1359 | 1359 | 1358 | 4076
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (8.3) | 64.6 (8.2) | 64.7 (8.2) | 64.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 419 | 442 | 483 | 1344
  Male | 940 | 917 | 875 | 2732
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 8 | 8 | 27
  Asian | 98 | 87 | 82 | 267
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 2 | 3
  Black or African American | 50 | 38 | 55 | 143
  White | 1162 | 1192 | 1180 | 3534
  More than one race | 4 | 9 | 5 | 18
  Unknown or Not Reported | 34 | 24 | 26 | 84
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram meter per square (kg/m^2)] — Population: Here, 'number analyzed' = participants with available data for the specified baseline measure.
  kilogram meter per square (kg/m^2)
    number analyzed (Participants) | 1359 | 1357 | 1357 | 4073
    (all) | 32.40 (6.01) | 32.81 (6.22) | 32.90 (6.21) | 32.70 (6.15)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurrence of Major Adverse Cardiovascular Events (MACE): Event Rate Per 100 Participant-years for First Occurrence of Major Cardiovascular (CV) Event - Non-Inferiority Analysis
Description: All MACE positively adjudicated by the clinical endpoint committee (CEC) were used in the analysis of the composite outcome of first occurrence to CV death, non-fatal myocardial infarction (MI), and non-fatal stroke. Kaplan-Meier curves of the cumulative event rate by treatment groups were used to depict the first occurrence of MACE over time. The event rate per 100 participant-years (calculated by 100*number of participants with events/sum of time at risk (days) over all participants/365.25) measured in terms of number of events per 100 participant-years was reported.
Time Frame: From Day 1 until the date of first adjudicated and confirmed occurrence of major CV event (maximum duration: up to 31.5 months)
Population: Analysis was performed on intent-to-treat (ITT) population. Data for this outcome measure (OM) was planned to be collected and analyzed for pooled population of participants who received Efpeglenatide (at any dose: 4 mg and 6 mg) as pre-specified in the protocol.
Measure: Number (95% Confidence Interval); unit: events per 100 participant-years
Groups:
- Efpeglenatide 4 mg+6 mg: Included all participants who received either Efpeglenatide 4 mg or 6 mg as SC injection once weekly up to end of treatment (median duration: 19.9 months).
Arm/Group | Efpeglenatide 4 mg+6 mg | Placebo
Number analyzed (Participants) | 2717 | 1359
events per 100 participant-years | 3.9 [3.4 to 4.5] | 5.3 [4.4 to 6.3]
Statistical Analysis 1: Comparison: Efpeglenatide 4 mg+6 mg vs Placebo; Hazard ratio and 95% Confidence Interval (CI) were obtained from a Cox proportional hazards model with region (North America, Latin America, Europe, other), randomization stratum of SGLT2 inhibitor use (current use, potential future use, neither current nor potential future use) and treatment (efpeglenatide 4 mg, efpeglenatide 6 mg, placebo) as fixed effect factor; Test type: Non-Inferiority — Non-inferiority of efpeglenatide 4 mg+6 mg versus placebo was to be claimed if the upper bound of the 2-sided 95% CI of the hazard ratio for the incidence of both 1.8 and less and 1.3 or less; p < .0001, Log Rank — One-sided p-value based on log rank test of hazard ratio for the incidence of both 1.8 and less and 1.3 or less; Hazard Ratio (HR) = 0.732, 95% CI 2-sided [0.583 to 0.918]

2. Secondary Outcome: Time to First Occurrence of Major Adverse Cardiovascular Events: Event Rate Per 100 Participant-years for First Occurrence of Major Cardiovascular Event - Superiority Analysis
Description: All MACE positively adjudicated by the CEC were used in the analysis of the composite outcome of first occurrence to CV death, non-fatal MI, and non-fatal stroke. Kaplan-Meier curves of the cumulative event rate by treatment groups were used to depict the first occurrence of MACE over time. The event rate per 100 participant-years (calculated by 100*number of participants with events/sum of time at risk (days) over all participants/365.25) measured in terms of number of events per 100 participant-years was reported.
Time Frame: as for outcome 1
Population: Analysis was performed on ITT population. Data for this OM was planned to be collected and analyzed for pooled population of participants who received Efpeglenatide (at any dose: 4 mg and 6 mg) as pre-specified in the protocol.
Measure: Number (95% Confidence Interval); unit: events per 100 participant-years
Arm/Group | Efpeglenatide 4 mg+6 mg | Placebo
Number analyzed (Participants) | 2717 | 1359
events per 100 participant-years | 3.9 [3.4 to 4.5] | 5.3 [4.4 to 6.3]
Statistical Analysis 1: Comparison: Efpeglenatide 4 mg+6 mg vs Placebo; Hazard ratio and 95% CI were obtained from a Cox proportional hazards model with region (North America, Latin America, Europe, other), randomization stratum of SGLT2 inhibitor use (current use, potential future use, neither current nor potential future use) and treatment (efpeglenatide 4 mg, efpeglenatide 6 mg, placebo) as fixed effect factor; Test type: Superiority — Superiority was claimed when the upper bound of the 2-sided 95% CI of hazard ratio was less than 1; p = 0.0069, Log Rank — Two-sided p-values based on log rank test of hazard ratio; Hazard Ratio (HR) = 0.732, 95% CI 2-sided [0.583 to 0.918]

3. Secondary Outcome: Time to First Occurrence of the Expanded Major Adverse Cardiovascular Events Composite Events: Event Rate Per 100 Participant-years for First Occurrence of Expanded Major Cardiovascular Event
Description: All MACE positively adjudicated by the CEC were used in the analysis of the expanded outcome of first occurrence to CV death (including fatal MI and fatal stroke), non-fatal MI, non-fatal stroke, coronary revascularization or hospitalization for unstable angina. Kaplan-Meier curves of the cumulative event rate by treatment groups were used to depict the first occurrence of MACE over time. The event rate per 100 participant-years (calculated by 100*number of participants with events/sum of time at risk (days) over all participants/365.25) measured in terms of number of events per 100 participant-years was reported. Data analysis was also performed independently by external steering committee for the publication.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: events per 100 participant-years
Arm/Group | Efpeglenatide 4 mg+6 mg | Placebo
Number analyzed (Participants) | 2717 | 1359
events per 100 participant-years | 5.4 | 6.8
Statistical Analysis 1: Comparison: Efpeglenatide 4 mg+6 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Superiority was claimed when the upper bound of the 2-sided 95% CI of hazard ratio was less than 1; p = 0.02, Log Rank — Two-sided p-values based on log rank test of hazard ratio; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.65 to 0.96]

4. Secondary Outcome: Time to First Occurrence of Composite Renal Endpoint: Event Rate Per 100 Participant-years for First Occurrence of Composite Renal Endpoint
Description: Composite renal endpoint included the following: incident macroalbuminuria (defined as urinary albumin-to-creatinine ratio of greater than (>) 300, as measured in mg of albumin to grams of creatinine, or >33.9, as measured in mg of albumin to millimoles of creatinine), plus an increase in urinary albumin-to-creatinine ratio of at least 30% from baseline, a sustained decrease in estimated glomerular filtration rate (eGFR) of at least 40% for 30 days or more, renal-replacement therapy for 90 days or more, and a sustained eGFR of less than 15 ml per minute per 1.73 m^2 for 30 days or more. Kaplan-Meier curves of the cumulative event rate by treatment groups were used to depict the first occurrence of renal endpoint over time. The event rate per 100 participant-years (calculated by 100*number of participants with events/sum of time at risk (days) over all participants/365.25) measured in terms of number of events per 100 participant-years was reported.
Time Frame: From Day 1 until the confirmed occurrence of composite renal endpoint (maximum duration: up to 31.5 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: events per 100 participant-years
Arm/Group | Efpeglenatide 4 mg+6 mg | Placebo
Number analyzed (Participants) | 2717 | 1359
events per 100 participant-years | 7.7 [6.9 to 8.6] | 11.6 [10.2 to 13.1]
Statistical Analysis 1: Comparison: Efpeglenatide 4 mg+6 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Superiority was claimed when the upper bound of the 2-sided 95% CI of hazard ratio was less than 1; p < .0001, Log Rank — Two-sided p-values based on log rank test of hazard ratio; Hazard Ratio (HR) = 0.675, 95% CI 2-sided [0.574 to 0.794]

ADVERSE EVENTS:
Time Frame: From time of first injection of investigational medicinal product (IMP) to the last injection of IMP + 30 days (i.e., up to maximum duration of 31.5 months).
Description: Reported adverse events (AEs) and deaths were treatment-emergent AEs (TEAEs), which was defined as AEs that developed/worsened/became serious during the TEAE period (defined as time from first injection of IMP to the last injection of IMP + 30 days). Safety population: all randomized participants who had received at least 1 dose of double-blind treatment, regardless of the amount of treatment administered, analyzed according to treatment actually received.
Arm/Group | Placebo | Efpeglenatide 4 mg | Efpeglenatide 6 mg
All-Cause Mortality (participants affected / at risk) | 49/1355 | 40/1360 | 25/1358
Serious Adverse Events (participants affected / at risk) | 298/1355 | 312/1360 | 275/1358
Other Adverse Events (participants affected / at risk) | 151/1355 | 348/1360 | 342/1358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1355) | Efpeglenatide 4 mg (N=1360) | Efpeglenatide 6 mg (N=1358)
Acquired Haemophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 2 (2)
Anaemia Vitamin B12 Deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypochromic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Left Ventricular Failure (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2)
Angina Pectoris (Cardiac disorders) | 10 (13) | 8 (8) | 17 (17)
Angina Unstable (Cardiac disorders) | 23 (29) | 20 (23) | 10 (11)
Aortic Valve Stenosis (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Arrhythmia Supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 12 (16) | 15 (17) | 12 (13)
Atrial Flutter (Cardiac disorders) | 2 (2) | 2 (2) | 5 (6)
Atrial Tachycardia (Cardiac disorders) | 1 (3) | 1 (1) | 0 (0)
Atrioventricular Block (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 4 (4) | 1 (1) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bundle Branch Block Left (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 5 (5) | 2 (2) | 1 (1)
Cardiac Discomfort (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 12 (12) | 4 (4) | 1 (1)
Cardiac Failure Acute (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Cardiac Failure Chronic (Cardiac disorders) | 2 (2) | 4 (4) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 3 (3) | 2 (2) | 2 (2)
Cardiac Valve Disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy Acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiovascular Insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 10 (11) | 14 (14) | 5 (5)
Coronary Artery Occlusion (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
Coronary Artery Stenosis (Cardiac disorders) | 1 (1) | 3 (3) | 3 (3)
Left Ventricular Dysfunction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Left Ventricular Failure (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 9 (10) | 4 (4) | 6 (6)
Myocardial Ischaemia (Cardiac disorders) | 4 (4) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus Node Dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 3 (4)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Tricuspid Valve Incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 3 (3) | 3 (4) | 2 (2)
Hypertrophic Cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Deafness Neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness Unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Meniere's Disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vestibular Disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Thyroid Mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroiditis Chronic (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Eyelid Ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Open Angle Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal Artery Embolism (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Incarcerated Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (6)
Colitis Ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal Sphincter Insufficiency (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Intestinal Ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mechanical Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mesenteric Artery Stenosis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obstructive Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Oesophageal Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Palatal Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2)
Pancreatitis Chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peptic Ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Varices Oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Accidental Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1) | 3 (3)
Cardiac Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 2 (2) | 0 (0)
Death (General disorders) | 4 (4) | 5 (5) | 4 (4)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired Healing (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 2 (2) | 6 (6) | 5 (5)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden Cardiac Death (General disorders) | 2 (2) | 5 (5) | 2 (2)
Sudden Death (General disorders) | 1 (1) | 2 (2) | 1 (1)
Vascular Stent Stenosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular Stent Thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 4 (4) | 3 (3)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 4 (4) | 3 (3)
Cholecystitis Chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (2) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic Cyst (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperplastic Cholecystopathy (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess Soft Tissue (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Arthritis Bacterial (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Atypical Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Bronchitis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 5 (5) | 1 (1) | 5 (5)
Covid-19 Pneumonia (Infections and infestations) | 5 (5) | 7 (7) | 6 (6)
Campylobacter Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 6 (7) | 3 (3) | 2 (4)
Cholangitis Infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Chronic Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Dermatitis Infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diabetic Foot Infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Diabetic Gangrene (Infections and infestations) | 2 (4) | 1 (2) | 1 (2)
Disseminated Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Enterococcal Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 6 (7)
Gastroenteritis Salmonella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Groin Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
H1n1 Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes Zoster Infection Neurological (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Joint Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Klebsiella Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Large Intestine Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised Infection (Infections and infestations) | 4 (7) | 2 (2) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oesophageal Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 5 (5) | 2 (2) | 3 (3)
Peritonitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pilonidal Cyst (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 15 (16) | 14 (14) | 9 (9)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 5 (5) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pyelonephritis Chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Renal Cyst Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Salpingitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Scrub Typhus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 9 (9) | 4 (4) | 4 (4)
Septic Shock (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Suspected Covid-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis Gastrointestinal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 7 (7) | 2 (5)
Urinary Tract Infection Enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Vulval Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Anastomotic Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Arterial Bypass Occlusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Arterial Bypass Stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Brachial Plexus Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 4 (4)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 3 (3)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Heat Exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Neck Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Patella Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Postoperative Respiratory Failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural Site Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Road Traffic Accident (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
Scapula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Stomal Hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Vascular Graft Thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anticoagulation Drug Level Above Therapeutic (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Glucose Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood Pressure Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Heart Rate Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lipase Increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Liver Function Test Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Plasminogen Activator Inhibitor Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Troponin Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 6 (6)
Diabetes Mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (3)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 2 (2)
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Food Intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (7) | 8 (9) | 2 (2)
Hyperglycaemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 8 (8) | 4 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lactic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Meniscal Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (4) | 2 (2)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 3 (3)
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Benign Neoplasm Of Scrotum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign Neoplasm Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Colorectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cutaneous T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Diffuse Large B-Cell Lymphoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0)
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine Tumour Of The Lung Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Non-Small Cell Lung Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal Adenocarcinoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 3 (3)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rectosigmoid Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Renal Cell Carcinoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Renal Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Spinal Cord Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous Cell Carcinoma Of The Oral Cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brain Injury (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid Artery Disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 2 (2) | 3 (3) | 4 (6)
Carotid Sinus Syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Cerebrovascular Disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular Insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cervicobrachial Syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic Hyperosmolar Coma (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (3) | 0 (0)
Facial Paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic Encephalopathy (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Hypoglycaemic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemic Unconsciousness (Nervous system disorders) | 4 (4) | 2 (2) | 2 (2)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Lacunar Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbosacral Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myasthenia Gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Senile Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 4 (5) | 7 (7)
Toxic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 3 (3) | 4 (4) | 2 (3)
Vith Nerve Paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vocal Cord Paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Device Fastener Issue (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Device Lead Issue (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Device Loosening (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Panic Attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 9 (9) | 10 (10) | 10 (11)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Diabetic Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Nephropathy Toxic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Tubulointerstitial Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary Bladder Polyp (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 2 (2)
Cervical Polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2)
Prostatic Atrophy (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 4 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleurocutaneous Fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 8 (9) | 8 (8) | 4 (4)
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 1 (1)
Aortic Stenosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Arterial Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Diabetic Vascular Disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Gangrene (Vascular disorders) | 2 (3) | 0 (0) | 0 (0)
Essential Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Extremity Necrosis (Vascular disorders) | 2 (2) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 2 (2)
Hypertensive Crisis (Vascular disorders) | 4 (4) | 4 (4) | 3 (3)
Hypertensive Emergency (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 4 (4) | 2 (2)
Intermittent Claudication (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 8 (8) | 7 (8) | 10 (10)
Peripheral Artery Occlusion (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral Artery Stenosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral Artery Thrombosis (Vascular disorders) | 0 (0) | 2 (3) | 0 (0)
Peripheral Circulatory Failure (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 3 (3) | 1 (1) | 2 (3)
Peripheral Vascular Disorder (Vascular disorders) | 5 (5) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous Thrombosis Limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1355) | Efpeglenatide 4 mg (N=1360) | Efpeglenatide 6 mg (N=1358)
Diarrhoea (Gastrointestinal disorders) | 64 (69) | 116 (139) | 117 (153)
Nausea (Gastrointestinal disorders) | 51 (60) | 196 (282) | 167 (194)
Vomiting (Gastrointestinal disorders) | 18 (19) | 85 (106) | 75 (95)
Decreased Appetite (Metabolism and nutrition disorders) | 15 (16) | 68 (74) | 77 (80)
Hypoglycaemia (Metabolism and nutrition disorders) | 37 (81) | 73 (159) | 53 (97)

LIMITATIONS AND CAVEATS:
The study was terminated early by the Sponsor but not due to any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT03496298/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT03496298/SAP_001.pdf